CLINICAL TRIAL: NCT00827853
Title: PolarCath® Cryoplasty Versus Conventional Balloon Post-dilation of Nitinol Stents for Peripheral Vascular Interventions (COBRA)
Brief Title: Study Comparing Two Methods of Expanding Stents Placed in Legs of Diabetics With Peripheral Vascular Disease
Acronym: COBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Subhash Banerjee, Chief of Cardiology, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOSTON SCI R&E 9-21-07#2
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: PERIPHERAL VASCULAR DISEASE
Keywords: Diabetes; Peripheral Vascular Disease (PVD); Superficial Femoral Artery (SFA); Cryoplasty; Restenosis
MeSH Terms: conditions — Peripheral Vascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Conventional angioplasty balloon post-dilation of nitinol self expanding stents
  Interventions: Procedure: Conventional angioplasty balloon
- 2 (Experimental): Cryoplasty balloon post-dilation
  Interventions: Procedure: cryoplasty balloon

INTERVENTIONS:
Procedure: Conventional angioplasty balloon — Post-dilation of clinically indicated nitinol self-expanding stents in the SFA using conventional angioplasty balloon
  Arms: 1
Procedure: cryoplasty balloon — Post-dilation of clinically indicated nitinol self-expanding stents in the SFA using cryoplasty balloon
  Arms: 2

SUMMARY:
Despite recent advances in stent technology and its widespread application in the treatment of peripheral vascular disease (PVD), incidences of partial or complete blockage of stent lumen (in-stent restenosis) due to in growth of cells (neo-intimal proliferation) is unacceptably high.

In diabetics with long superficial femoral artery (SFA) lesions, in-stent restenosis rates are higher than in non-diabetics. Consequently interventional techniques that curtail in-stent restenosis have to be explored. Cryoplasty is a stent expansion method in which a balloon is expanded using pressurized nitrous oxide gas. As the nitrous oxide expands in the balloon it cools the surroundings to about -10 degrees C. This induces programed death (apoptosis) of the smooth muscle cells in arterial wall.

The investigators hypothesize that Cryoplasty, by inducing an apoptotic smooth muscle cell response, when applied to post-dilation of nitinol self-expanding stents in the Superficial Femoral Artery (SFA) of diabetics, would lead to decreased in-stent restenosis due to decreased neointimal proliferation.

DETAILED DESCRIPTION:
The pre-recruitment process would identify diabetics who have life-style limiting claudication in their legs. Based on the physicians decision such patients may have to undergo a peripheral vascular intervention of the SFA, with placement of self-expanding nitinol stents. If such a decision is made, the patient will be randomized to either cryoplasty balloon post-dilation of the stent or to conventional angioplasty balloon post-dilation after obtaining informed consent. At one year, in segment (stent + 10 mm beyond its proximal and distal edges) peak systolic velocity by duplex ultrasound will be measured in all subjects to assess the rate of binary restenosis defined as a > or = 2.5 times increase in peak systolic velocity (primary endpoint). A 6 month resting ankle brachial index, and binary restenosis may be assessed as a secondary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics, insulin or non-insulin dependent above 21 years of age
* Able to provide an informed consent
* Life expectancy > 1 year
* Presenting with with moderate claudication (Rutherford stage 2), severe intermittent claudication (Rutherford stage 3), chronic critical limb ischemia with pain while the patient was at rest(Rutherford stage 4), or chronic critical limb ischemia with ischemic ulcers/gangrene(Rutherford stage 5/6)
* Placement of > 5 mm in diameter self-expanding Nitinol stent in the SFA, with at least 1 vessel infra-popliteal runoff
* Placement of > 60 mm in length self-expanding Nitinol stent in the SFA, with at least 1 vessel infra-popliteal runoff

Exclusion Criteria:

* Serum creatinine of >= 2.0 mg/dl
* Presence of iodinated contrast allergy
* Presence of allergy to Aspirin and Plavix
* Pregnancy
* Relative or absolute contraindication for anticoagulation
* History of allergy to Angiomax and unfractionated heparin or heparin induced thrombocytopenia (HIT)
* White blood count < 3000; platelet count < 100000, and baseline hemoglobin < 10 g/dl
* Absence of brisk at least 1 vessel infra-popliteal runoff to the foot
* Left ventricular ejection fraction < 25%
* Relative or absolute contraindication for anticoagulation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Rate of binary restenosis as determined by duplex ultrasound. | 1 year

SECONDARY OUTCOMES:
Resting ankle-brachial index | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — VA North Texas Healthcare Systen, Dallas, TX; Emmanouil S Brilakis, MD, PhD, Study Director — VA North Texas Healtcare System, Dallas, TX; Tony S Das, MD, Study Director — Texas Health Resources
Locations (4):
- United States (4):
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - VA Medical Center, Oklahoma City, Oklahoma
  - Dallas Veterans Hospital, Dallas, Texas
  - Dallas Presbyterian Hospital, Dallas, Texas

REFERENCES:
- [Background] Minar E, Pokrajac B, Maca T, Ahmadi R, Fellner C, Mittlbock M, Seitz W, Wolfram R, Potter R. Endovascular brachytherapy for prophylaxis of restenosis after femoropopliteal angioplasty : results of a prospective randomized study. Circulation. 2000 Nov 28;102(22):2694-9. doi: 10.1161/01.cir.102.22.2694. PMID 11094034
- [Background] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699
- [Background] Cejna M, Thurnher S, Illiasch H, Horvath W, Waldenberger P, Hornik K, Lammer J. PTA versus Palmaz stent placement in femoropopliteal artery obstructions: a multicenter prospective randomized study. J Vasc Interv Radiol. 2001 Jan;12(1):23-31. doi: 10.1016/s1051-0443(07)61397-9. PMID 11200349
- [Background] Becquemin JP, Favre JP, Marzelle J, Nemoz C, Corsin C, Leizorovicz A. Systematic versus selective stent placement after superficial femoral artery balloon angioplasty: a multicenter prospective randomized study. J Vasc Surg. 2003 Mar;37(3):487-94. doi: 10.1067/mva.2003.155. PMID 12618680
- [Background] Sabeti S, Mlekusch W, Amighi J, Minar E, Schillinger M. Primary patency of long-segment self-expanding nitinol stents in the femoropopliteal arteries. J Endovasc Ther. 2005 Feb;12(1):6-12. doi: 10.1583/04-1359.1. PMID 15683273
- [Background] Johnston KW. Femoral and popliteal arteries: reanalysis of results of balloon angioplasty. Radiology. 1992 Jun;183(3):767-71. doi: 10.1148/radiology.183.3.1294068.
- [Background] Zdanowski Z, Albrechtsson U, Lundin A, Jonung T, Ribbe E, Thorne J, Norgren L. Percutaneous transluminal angioplasty with or without stenting for femoropopliteal occlusions? A randomized controlled study. Int Angiol. 1999 Dec;18(4):251-5. PMID 10811511
- [Background] Sabeti S, Schillinger M, Amighi J, Sherif C, Mlekusch W, Ahmadi R, Minar E. Primary patency of femoropopliteal arteries treated with nitinol versus stainless steel self-expanding stents: propensity score-adjusted analysis. Radiology. 2004 Aug;232(2):516-21. doi: 10.1148/radiol.2322031345. PMID 15286322
- [Background] Duda SH, Pusich B, Richter G, Landwehr P, Oliva VL, Tielbeek A, Wiesinger B, Hak JB, Tielemans H, Ziemer G, Cristea E, Lansky A, Beregi JP. Sirolimus-eluting stents for the treatment of obstructive superficial femoral artery disease: six-month results. Circulation. 2002 Sep 17;106(12):1505-9. doi: 10.1161/01.cir.0000029746.10018.36. PMID 12234956
- [Background] Schillinger M, Exner M, Mlekusch W, Haumer M, Sabeti S, Ahmadi R, Schwarzinger I, Wagner O, Minar E. Restenosis after femoropopliteal PTA and elective stent implantation: predictive value of monocyte counts. J Endovasc Ther. 2003 Jun;10(3):557-65. doi: 10.1177/152660280301000322. PMID 12932168
- [Background] Yiu WK, Cheng SW, Sumpio BE. Vascular smooth muscle cell apoptosis induced by "supercooling" and rewarming. J Vasc Interv Radiol. 2006 Dec;17(12):1971-7. doi: 10.1097/01.RVI.0000244868.65867.FB. PMID 17185696
- [Background] Venkatasubramanian RT, Grassl ED, Barocas VH, Lafontaine D, Bischof JC. Effects of freezing and cryopreservation on the mechanical properties of arteries. Ann Biomed Eng. 2006 May;34(5):823-32. doi: 10.1007/s10439-005-9044-x. Epub 2006 Apr 18. PMID 16619131
- [Background] Grassl ED, Bischof JC. In vitro model systems for evaluation of smooth muscle cell response to cryoplasty. Cryobiology. 2005 Apr;50(2):162-73. doi: 10.1016/j.cryobiol.2005.01.002. PMID 15843006
- [Background] Laird J, Jaff MR, Biamino G, McNamara T, Scheinert D, Zetterlund P, Moen E, Joye JD. Cryoplasty for the treatment of femoropopliteal arterial disease: results of a prospective, multicenter registry. J Vasc Interv Radiol. 2005 Aug;16(8):1067-73. doi: 10.1097/01.RVI.0000167866.86201.4E. PMID 16105918
- [Derived] Banerjee S, Das TS, Abu-Fadel MS, Dippel EJ, Shammas NW, Tran DL, Zankar A, Varghese C, Kelly KC, Weideman RA, Little BB, Reilly RF, Addo T, Brilakis ES. Pilot trial of cryoplasty or conventional balloon post-dilation of nitinol stents for revascularization of peripheral arterial segments: the COBRA trial. J Am Coll Cardiol. 2012 Oct 9;60(15):1352-9. doi: 10.1016/j.jacc.2012.05.042. Epub 2012 Sep 12. PMID 22981558